CLINICAL TRIAL: NCT02816593
Title: In-office and At-home Tooth Bleaching Using Low Concentration Peroxides.: Effectiveness, Security and Impact on Quality of Life Related to Oral Health
Brief Title: In-office and At-home Tooth Bleaching Using Low Concentration Peroxides.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Cláudia Silami de Magalhães, Associate Professor IV, Department of Restorative Dentistry at the Federal University of Minas Gerais, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUMinasGerais01
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Discolored Teeth
Keywords: carbamide peroxide; Hydrogen peroxide; Quality of life
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 - HP 6% (Experimental): Group 1: Experimental: Office; hydrogen peroxide 6%,
  Interventions: Drug: hydrogen peroxide 6%
- Group 2 - HP 15% (Experimental): Group 2: Experimental: Office; hydrogen peroxide 15%,
  Interventions: Drug: hydrogen peroxide 15%
- Group 3 - CP 10% (Active Comparator): Group 3: Control: Homemade; Carbamide Peroxide 10%,
  Interventions: Drug: Carbamide Peroxide 10%

INTERVENTIONS:
Drug: hydrogen peroxide 6% — Office; hydrogen peroxide 6%, 3 sessions of 20 minutes of application
  Other Names: Group 1 - HP 6%
  Arms: Group 1 - HP 6%
Drug: hydrogen peroxide 15% — Office; hydrogen peroxide 15%, 3 sessions of 20 minutes of application
  Other Names: Group 2 - HP 15%
  Arms: Group 2 - HP 15%
Drug: Carbamide Peroxide 10% — Homemade; Carbamide Peroxide 10%, 2 hours per day for 21 days
  Other Names: Group 3 - CP 10%
  Arms: Group 3 - CP 10%

SUMMARY:
To evaluate the efficacy, safety and impact on quality of life related to oral health of home and office tooth whitening techniques in young individuals.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy, safety and impact on quality of life related to oral health of tooth whitening techniques in young individuals. It will be a randomized, parallel and single blind. Participants are divided into three groups (n = 30) according to bleaching technique to be performed (G1 = Office / hydrogen peroxide 6%; G2 = Office / hydrogen peroxide 15%; G3 = Home / carbamide peroxide 10%). The color of the teeth will be evaluated in seven different times, using the color scale Vita Master Classic 3D and spectrophotometer Vita Easy Shade Advance. IGM (1986) - the presence of tooth sensitivity by visual analogue scale and gingival security through modified gingival index will be evaluated. The impact of bleaching quality of life will be assessed using the Brazilian version of the oral impact on daily performance (OIDP). The instrument will be applied in interview form at two different times at baseline (T0) and thirty days after the first evaluation (T4). Statistical analysis include descriptive analysis and testing to compare the two bleaching techniques as the color change, sensitivity, gum irritation and impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* tooth color ranging from A3 or darker, teeth with no stains and restorations without whitening experience

Exclusion Criteria:

* participants with gingivitis and periodontal disease, the total biofilm accumulation greater than 30%, severe crowding dental, smoking with tooth sensitivity and pregnant women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of color change | T0 (Baseline): Before treatment;T1:After one week of starting treatment;T2: After 2 weeks of starting treatment;T3: After 3 weeks of starting treatment;T4: After 30 days of starting treatment;T5:After 6 months ;T6:After 12 months
  Visual evaluation using color scale Vita Classical 3D Master (Vita Zahnfabrik, Germany); (B1, A1, B2, D2, A2, C1, C2, D4, A3, D3, B3, A3.5, B4, C3, A4, C4) Quantitative evaluation using a spectrophotometer Easy Shade Advance ® (Wilcos Brazil).
  System CIE L * a * b * - L represents the value (lightness or darkness), the value of a * is a measure red (positive a *) or green (negative a *); the value of b * is a yellow extent (b * positive) or blue (b * negative) and the color difference between the color coordinate is calculated as ΔE * = [(ΔL *) 2 + (Δa *) 2 + (Δb *) 2] 1/2.

SECONDARY OUTCOMES:
Tooth sensitivity assessment | T0 (Baseline): Before treatment;T1:After one week of starting treatment;T2: After 2 weeks of starting treatment;T3: After 3 weeks of starting treatment;T4: After 30 days of starting treatment;
  It will be registered according to the Visual Analogue Scale (VAS), according to the criteria: none, mild, moderate or severe.
Evaluation of gingival irritation | T0 (Baseline): Before treatment;T1:After one week of starting treatment;T2: After 2 weeks of starting treatment;T3: After 3 weeks of starting treatment;T4: After 30 days of starting treatment;
  The Modified Gingival Index (IGM) The criteria are as follows: 0: Absence of inflammation;1: mild inflammation - slight change in color and texture of the gum; 2: mild inflammation involving the entire gingival margin; 3: moderate inflammation, shiny surface and edema; 4: Severe inflammation, spontaneous bleeding and severe edema.
Impact assessment on quality of life | T0 (Baseline): Before treatment;T4: After 30 days of starting treatment;
  The Brazilian version of the oral impact on daily performance (OIDP) will be used to assess the impact on quality of life. The instrument will be applied in interview form at two different times at baseline (T0) and thirty days after the first evaluation (T4) to assess the perception of changes in oral health after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nayara Kelly Lyrio Ferraz, Principal Investigator — PhD student of Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin J, Vildosola P, Bersezio C, Herrera A, Bortolatto J, Saad JR, Oliveira OB Jr, Fernandez E. Effectiveness of 6% hydrogen peroxide concentration for tooth bleaching-A double-blind, randomized clinical trial. J Dent. 2015 Aug;43(8):965-72. doi: 10.1016/j.jdent.2015.05.011. Epub 2015 Jun 6. PMID 26057085
- [Background] Meireles SS, Goettems ML, Dantas RV, Bona AD, Santos IS, Demarco FF. Changes in oral health related quality of life after dental bleaching in a double-blind randomized clinical trial. J Dent. 2014 Feb;42(2):114-21. doi: 10.1016/j.jdent.2013.11.022. Epub 2013 Dec 4. PMID 24316342